CLINICAL TRIAL: NCT03688308
Title: Randomized Control Trial of Bone Marrow Derived Stem Cells Combined With Arthroscopic Surgery Versus Arthroscopic Surgery Only for the Treatment of Rotator Cuff Tears
Brief Title: Bone Marrow Derived Stem Cells for the Treatment of Rotator Cuff Tears
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in personnel
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-47762
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Injury
Keywords: Bone marrow aspirate; Biologics
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not know if they received the surgical intervention that includes BMAC administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder arthroscopy with BMAC (Experimental): This arm will have patients who receive surgical intervention with arthroscopic rotator cuff repair along with 3-4cc of BMAC produced from the Harvest/Terumo BCT system
  Interventions: Procedure: Arthroscopic rotator cuff repair with bone marrow aspirate concentrate
- Shoulder arthroscopy alone (Active Comparator): This arm will have patients who receive surgical intervention with arthroscopic rotator cuff repair without administration of BMAC.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair with bone marrow aspirate concentrate — Subjects will undergo shoulder arthroscopy for rotator cuff repair using a double row technique. Subjects will also be injected with bone marrow aspirate concentrate harvested from the pelvis and centrifuged prior to injection in the shoulder (produced using the Harvest/Terumo BCT system)
  Other Names: Injection of bone marrow aspirate concentrate harvested from the patient's iliac crest (produced using the Harvest/Terumo BCT system)
  Arms: Shoulder arthroscopy with BMAC
Procedure: Arthroscopic rotator cuff repair — Subjects will undergo shoulder arthroscopy for rotator cuff repair using a double row technique.
  Arms: Shoulder arthroscopy alone

SUMMARY:
The primary objective is to determine whether adjunct treatment using bone marrow aspirate concentrate (BMAC) in conjunction with arthroscopic repair of rotator cuff tears reduces retear rates compared to a control population undergoing arthroscopic repair without BMAC administration. The secondary objectives are to (1) evaluate the survival and incorporation of BMAC labeled cells with MRI imaging using the Ferumoxytol infusion stem cell labeling technique, and (2) determine if administration of BMAC leads to better clinical outcomes as measured by ASES, UCLA and Constant scoring metrics.

DETAILED DESCRIPTION:
Rotator cuff repair and regeneration has become a focal point for scientists and surgeons in search for a biological treatment to improve tendon healing, especially in situations of unfavorable biological conditions. Recent literature supports harvesting and centrifuging bone marrow aspirate to produce bone marrow aspirate concentration (BMAC) in hopes that mesenchymal stem cells in the bone marrow aspirate can promote tendon healing and regeneration.

This is a single blinded randomized clinical trial using labeled BMAC cells in adults diagnosed with medium to large, single tears of the rotator cuff. This is a single site study where at least 45 cases among eligible patients will be identified and randomly assigned to a either a control (arthroscopic repair without BMAC) group or experimental (arthroscopic repair with BMAC) group. A power analysis will be performed after enrolling 20 patients to determine the total number of patients required to reach adequate power.

A patient will receive an infusion of Ferumoxytol 1 day prior to the surgical procedure. An infusion nurse will be present at all times during the infusion to monitor vitals. On the day of the surgical procedure patients in the both groups will undergo arthroscopic rotator cuff repair using a double-row technique. Patients in the experimental group will also undergo harvesting of bone marrow aspirate from the anterior inferior iliac crest, which will be centrifuged to about 3-4cc of BMAC and placed beneath the tendon at the bone interface. MRIs will be completed on days 1 and 7 post-operatively to track retention of the labeled mesenchymal cells. Ultrasound imaging will be performed at 6 months post-surgery to evaluate tendon healing. Final MRIs will be obtained at 1 year and 2 years post surgery. Patient related outcomes will be collected at the pre-operative visit, 3 months, 6 months, 1 year and 2 years post surgery in the forms of ASES, UCLA and Constant scoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50-75 patients with MRI confirmed rotator cuff tears sized 1.5-3cm including supraspinatus with or without an associated partial infraspinatus or subscapularis tear
* Chronic tear > 3 months
* Failed a minimum of 6 weeks of physical therapy
* Hamada stage 1
* Goutallier staging < 3

Exclusion Criteria:

* Radiographs demonstrating mild to moderate arthritis
* Diagnosis of Inflammatory (RA, JIA etc) or infectious arthritis
* Hamada stage > 2
* Cortisone and/or Hyaluronic acid intra-articular injection within the last 3 months
* Brachial plexus pathology
* Currently pregnant or planning to become pregnant
* Shoulder PRP injection within the last year
* History of iron overload syndrome
* Concurrent surgery for shoulder instability

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Tendon healing rates | 24 months
  Percent of rotator cuff repairs that demonstrate full healing at 2 years post surgery

SECONDARY OUTCOMES:
UCLA Score | Date of enrollment to 24 months post-operatively
  UCLA score (0-35 points; higher score is better) at 24 months post surgery to measure functional outcome.
ASES Score | Date of enrollment to 24 months post-operatively
  American Shoulder and Elbow Surgeons Shoulder Score (ASES) (0-100 points; higher score is better) at 24 months to measure functional outcome.
Constant Score | Date of enrollment to 24 months post-operatively
  Constant score (0-100 points; higher score is better) at 24 months.
Retention of the mesenchymal stem cells | 7 days
  Imaging of labeled mesenchymal stems cells in the shoulder to assess retention post injection

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Dragoo, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No